CLINICAL TRIAL: NCT05304104
Title: Building an Equitable and Accessible System of Eating Disorder Care for VA, DoD, and Underrepresented Americans With Eating Disorders (EASED Study)
Brief Title: Building an Equitable and Accessible System of Eating Disorder Care for VA, DoD, and Underrepresented Americans
Acronym: EASED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1645520; CDMRP-PR203460 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-02-18; First posted 2022-03-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Binge-Eating Disorder; Bulimia Nervosa; Veterans Health; Cognitive Behavioral Therapy
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Cognitive Behavioral Therapy (teleCBT) (Experimental): About one-half of participants will be randomly assigned to Telehealth Cognitive Behavioral Therapy (teleCBT), a virtual Cognitive Behavioral Therapy (CBT) for binge eating disorders delivered via an Office of Information and Technology (OI&T)-approved video platform, by a master's-level research clinician. TeleCBT will be administered in 8 to 10 hourly individual sessions over a three-month treatment period.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Self-Help Cognitive Behavioral Therapy (shCBT) (Active Comparator): About one-half of participants will be randomly assigned to Self-Help Cognitive Behavioral Therapy (shCBT), a Self-Help CBT for binge eating disorders initiated by a research assistant via telephone and then continued by the participant at home. These materials are the same exact ones provided to participants in TeleCBT (i.e., treatments are matched for materials), and will be mailed to participants. They will be instructed to work independently through one chapter per week for the following 12 weeks (i.e., treatment length is matched to TeleCBT).
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The treatment has three stages. Stage 1 consists of presentation of the CBT model; introduction and discussion of the structure, goals, interventions, and expected outcome of treatment; education regarding binge eating and dieting; and the introduction of self-monitoring techniques for identifying problematic eating practices and triggers. Stage 2 consists of maintaining the normalized eating and self-monitoring procedures but becomes increasingly cognitively oriented. Stage 3 focuses on practicing skills, consolidation of progress and relapse prevention. Treatment will adhere to a manual developed by Dr. Masheb (PI), adapted for Veterans, and written at a seventh-grade reading level.

SUMMARY:
When untreated, eating disorders present with tremendous burdens to affected active duty Service members and Veterans and their families, and are very costly to the DoD and VA healthcare system. A comparative effectiveness study with state-of-the-art virtual treatment for BN and BED specifically adapted for testing with the Veteran population and other underrepresented eating disorder populations will lead to major improvements in clinical outcomes. The treatment will be integrated with VA's newest telehealth technology to profoundly enhance access to care anywhere, at any time. This trial of therapist-led and self-help CBT treatments, combined with our expert panel methods to inform VA Clinical Practice Guidelines for Eating Disorders and plans for dissemination, will accelerate the pace for the transition of results both for large-scale deployment in the VA system and for real-world impact among diverse and underrepresented eating disorder populations.

DETAILED DESCRIPTION:
The overall objective is to test and improve access to evidence-based eating disorder treatment for active duty Service members and Veterans. The two-part project will include a comparative effectiveness trial of virtual treatments followed by qualitative methods for implementation. The randomized controlled trial will specifically test the effectiveness of Telehealth Cognitive Behavioral Therapy (TeleCBT) compared to Self-Help Cognitive Behavioral Therapy (shCBT) for binge eating disorders.

* Aim 1 (Superiority): To assess the effectiveness of TeleMental Health CBT (TeleCBT) compared to Self-Help CBT (shCBT) for decreasing binge frequency (primary) and improving eating behavior and mental health outcomes.

  1. It is hypothesized that Veterans in TeleCBT will have greater reductions in binge frequency, and greater percentage of participants who are binge remitted, than Veterans in shCBT.
  2. It is further hypothesized that TeleCBT will have better outcomes on purging behavior (among those with BN), eating pathology, symptoms of depression and trauma, and quality of life than shCBT.
* Aim 2 (Process): To assess demographic (age and gender) and clinical (clinical severity and comorbidity) characteristics as potential predictors, moderators and correlates of treatment outcome.
* Aim 3 (Implementation): To inform VA Clinical Practice Guidelines for Eating Disorders by convening a panel of experts and utilizing qualitative consensus building methods (Delphi Method) to develop evidence-based recommendations regarding dissemination and implementation of treatment for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Presence of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Bulimia Nervosa (BN) or Binge Eating Disorder (BED)
* Veteran Health Administration (VHA) user

Exclusion Criteria:

* Active psychosis or high acute risk for suicide
* Medical or psychiatric illness, or cognitive deficits, that interfere with providing consent, completing assessments, or engaging in treatment for eating disorders
* Pregnancy or lactation
* Patients with suspected Anorexia or Atypical Anorexia will be excluded and referred to other VA care services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in binge frequency as assessed by Eating Disorder Examination-Interview 17.0th Edition (EDE). | baseline, 3 months (post-treatment), and 6 months
  The EDE is the structured diagnostic interview that is considered the gold-standard to diagnose, and assess the symptoms of, eating disorders including binge eating, purging behaviors, and eating disorder pathology.
Change in Eating Disorder Examination-Self-report Questionnaire (EDE-Q) | baseline, 3 months (post-treatment), and 6 months
  The EDE-Q is the self-report version of the more intensive EDE interview. Research has documented that the EDE-Q performs well as a measure of change in treatment trials61and has adequate convergence with the interview format62,63. The EDE-Q generates the same frequency data for eating behaviors (binge eating and overeating) in the past 28 days, and the same four subscales reflecting eating disorder pathology.

SECONDARY OUTCOMES:
A change in depression score as assessed by the Patient Health Questionnaire-9 (PHQ-9). | baseline, 3 months (post-treatment), and 6 months
  The PHQ-9 a 9-item self-report questionnaire used to assess for the presence and severity of the symptoms of depression.
A change in post-traumatic stress disorder (PTSD) as assessed by the PTSD Checklist-5 (PCL-5) with Criterion A. | baseline, 3 months (post-treatment), and 6 months
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Criterion A will be assessed using a standard brief assessment.
Self-assessment of overall wellness as assessed by the Yale Eating and Weight Quality of Life Scale (Yale QoL) and the Visual Analog Scale (VAS) within the European Quality of Life Screener (Euro QoL). | baseline, 3 months (post-treatment), and 6 months
  Yale QoL evaluates eight aspects of overall quality of life based specifically on the impact of weight or eating on each domain (physical activity, self-care, daily responsibilities, relationships, public distress, physical discomfort, emotional distress, and shame or guilt). The VAS is used to assess perceived health status ranging from 0 to 100.
Participant engagement in treatment and treatment satisfaction as assessed by our own Skills Confidence , Materials Engagement, and Treatment Satisfaction surveys. | 3 months (post-treatment)
  The Skills Confidence survey is a 12-item measure used to determine a participant's level of confidence in a number of skills taught during treatment. Participants can answer on a scale ranging from strongly disagree to strongly agree. The Materials Engagement survey is an 11-item measure used to determine a participant's level of engagement in the materials. The Treatment Satisfaction survey is an 11-item measure that is used to determine how helpful a number of skills were to manage a participant's binge eating behaviors on a scale from 0 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Masheb, PhD, Principal Investigator — VA Connecticut Research Department
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agras WS, Fitzsimmons-Craft EE, Wilfley DE. Evolution of cognitive-behavioral therapy for eating disorders. Behav Res Ther. 2017 Jan;88:26-36. doi: 10.1016/j.brat.2016.09.004. PMID 28110674
- [Background] Allison KC, Lundgren JD, O'Reardon JP, Martino NS, Sarwer DB, Wadden TA, Crosby RD, Engel SG, Stunkard AJ. The Night Eating Questionnaire (NEQ): psychometric properties of a measure of severity of the Night Eating Syndrome. Eat Behav. 2008 Jan;9(1):62-72. doi: 10.1016/j.eatbeh.2007.03.007. Epub 2007 Mar 28. PMID 18167324
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Publishing; 2013.
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- [Background] Bartlett BA, Mitchell KS. Eating disorders in military and veteran men and women: A systematic review. Int J Eat Disord. 2015 Dec;48(8):1057-69. doi: 10.1002/eat.22454. Epub 2015 Aug 27. PMID 26310193
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Bellows BK, DuVall SL, Kamauu AW, Supina D, Babcock T, LaFleur J. Healthcare costs and resource utilization of patients with binge-eating disorder and eating disorder not otherwise specified in the Department of Veterans Affairs. Int J Eat Disord. 2015 Dec;48(8):1082-91. doi: 10.1002/eat.22427. Epub 2015 May 8. PMID 25959636
- [Background] Bellows BK, LaFleur J, Kamauu AW, Ginter T, Forbush TB, Agbor S, Supina D, Hodgkins P, DuVall SL. Automated identification of patients with a diagnosis of binge eating disorder from narrative electronic health records. J Am Med Inform Assoc. 2014 Feb;21(e1):e163-8. doi: 10.1136/amiajnl-2013-001859. Epub 2013 Nov 7. PMID 24201026
- [Background] Daeppen JB, Yersin B, Landry U, Pecoud A, Decrey H. Reliability and validity of the Alcohol Use Disorders Identification Test (AUDIT) imbedded within a general health risk screening questionnaire: results of a survey in 332 primary care patients. Alcohol Clin Exp Res. 2000 May;24(5):659-65. PMID 10832907
- [Background] Economic Research Service, USDA. U.S. Household Food Security Survey Module: Six-Item Short Form. 2012.
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Fairburn C, Cooper Z, O'Connor M. Eating disorder examination: Edition 17.0D. 2014.
- [Background] Fairburn, C. G. & cooper, Z. The eating disorder examination. in Fairburn, C. G., Wilson, G. T., & Schleimer, K. (1993). Binge eating: Nature, assessment, and treatment (pp. 317-360). New York: Guilford Press.
- [Background] Fairburn C. Overcoming binge eating. Guilford Press; 1995.
- [Background] Foa EB, Riggs DS, Dancu CV, Rothbaum BO. Reliability and validity of a brief instrument for assessing post-traumatic stress disorder. J Traum Stress. 1993;6(4):459-473. https://doi.org/10.1002/jts.2490060405. doi: https://doi.org/10.1002/jts.2490060405.
- [Background] Forbush KT, Wildes JE, Pollack LO, Dunbar D, Luo J, Patterson K, Petruzzi L, Pollpeter M, Miller H, Stone A, Bright A, Watson D. Development and validation of the Eating Pathology Symptoms Inventory (EPSI). Psychol Assess. 2013 Sep;25(3):859-78. doi: 10.1037/a0032639. Epub 2013 Jul 1. PMID 23815116
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Godin G. The godin-shephard leisure-time physical activity questionnaire. Health Fit J Can. 2011;4(1):18-22. https://hfjc.library.ubc.ca/index.php/HFJC/article/view/82. doi: 10.14288/hfjc.v4i1.82.
- [Background] Gratz, K. L. & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54.
- [Background] Grilo CM, Masheb RM, Brody M, Burke-Martindale CH, Rothschild BS. Binge eating and self-esteem predict body image dissatisfaction among obese men and women seeking bariatric surgery. Int J Eat Disord. 2005 May;37(4):347-51. doi: 10.1002/eat.20130. PMID 15856499
- [Background] Grilo CM, Masheb RM, Salant SL. Cognitive behavioral therapy guided self-help and orlistat for the treatment of binge eating disorder: a randomized, double-blind, placebo-controlled trial. Biol Psychiatry. 2005 May 15;57(10):1193-201. doi: 10.1016/j.biopsych.2005.03.001. PMID 15866560
- [Background] Grilo CM, Masheb RM, Wilson GT. A comparison of different methods for assessing the features of eating disorders in patients with binge eating disorder. J Consult Clin Psychol. 2001 Apr;69(2):317-22. doi: 10.1037//0022-006x.69.2.317. PMID 11393608
- [Background] Grilo CM, Masheb RM, Wilson GT, Gueorguieva R, White MA. Cognitive-behavioral therapy, behavioral weight loss, and sequential treatment for obese patients with binge-eating disorder: a randomized controlled trial. J Consult Clin Psychol. 2011 Oct;79(5):675-85. doi: 10.1037/a0025049. PMID 21859185
- [Background] Grilo CM, Masheb RM, Wilson GT. Different methods for assessing the features of eating disorders in patients with binge eating disorder: a replication. Obes Res. 2001 Jul;9(7):418-22. doi: 10.1038/oby.2001.55. PMID 11445665
- [Background] Grilo CM, Masheb RM, Wilson GT. Efficacy of cognitive behavioral therapy and fluoxetine for the treatment of binge eating disorder: a randomized double-blind placebo-controlled comparison. Biol Psychiatry. 2005 Feb 1;57(3):301-9. doi: 10.1016/j.biopsych.2004.11.002. PMID 15691532
- [Background] Guerdjikova AI, McElroy SL, Winstanley EL, Nelson EB, Mori N, McCoy J, Keck PE Jr, Hudson JI. Duloxetine in the treatment of binge eating disorder with depressive disorders: a placebo-controlled trial. Int J Eat Disord. 2012 Mar;45(2):281-9. doi: 10.1002/eat.20946. Epub 2011 Jul 8. PMID 21744377
- [Background] Gueorguieva R, Krystal JH. Move over ANOVA: progress in analyzing repeated-measures data and its reflection in papers published in the Archives of General Psychiatry. Arch Gen Psychiatry. 2004 Mar;61(3):310-7. doi: 10.1001/archpsyc.61.3.310. PMID 14993119
- [Background] Gusi, N., P. Olivares, and R. Rajendram, The EQ-5D Health-Related Quality of Life Questionnaire, in Handbook of Disease Burdens and Quality of Life Measures R.R.W. Victor R. Preedy, Editor. 2010, Springer New York: New York. p. 87-99.
- [Background] Hedeker D, Mermelstein RJ, Demirtas H. Analysis of binary outcomes with missing data: missing = smoking, last observation carried forward, and a little multiple imputation. Addiction. 2007 Oct;102(10):1564-73. doi: 10.1111/j.1360-0443.2007.01946.x. PMID 17854333
- [Background] Higgins DM, Dorflinger L, MacGregor KL, Heapy AA, Goulet JL, Ruser C. Binge eating behavior among a national sample of overweight and obese veterans. Obesity (Silver Spring). 2013 May;21(5):900-3. doi: 10.1002/oby.20160. PMID 23784891
- [Background] Hilbert A, Bishop ME, Stein RI, Tanofsky-Kraff M, Swenson AK, Welch RR, Wilfley DE. Long-term efficacy of psychological treatments for binge eating disorder. Br J Psychiatry. 2012 Mar;200(3):232-7. doi: 10.1192/bjp.bp.110.089664. Epub 2012 Jan 26. PMID 22282429
- [Background] Hilbert A, Petroff D, Herpertz S, Pietrowsky R, Tuschen-Caffier B, Vocks S, Schmidt R. Meta-analysis of the efficacy of psychological and medical treatments for binge-eating disorder. J Consult Clin Psychol. 2019 Jan;87(1):91-105. doi: 10.1037/ccp0000358. PMID 30570304
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems and barriers to care. US Army Med Dep J. 2008 Jul-Sep:7-17. PMID 20088060
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Kroenke K, Spitzer RL. The PHQ-9: A new depression diagnostic and severity measure. Psychiatric Annals. 2002;32(9):509-515. doi: 10.3928/0048-5713-20020901-06.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Latner JD, Mond JM, Kelly MC, Haynes SN, Hay PJ. The Loss of Control Over Eating Scale: development and psychometric evaluation. Int J Eat Disord. 2014 Sep;47(6):647-59. doi: 10.1002/eat.22296. Epub 2014 May 26. PMID 24862351
- [Background] Linardon J, Fairburn CG, Fitzsimmons-Craft EE, Wilfley DE, Brennan L. The empirical status of the third-wave behaviour therapies for the treatment of eating disorders: A systematic review. Clin Psychol Rev. 2017 Dec;58:125-140. doi: 10.1016/j.cpr.2017.10.005. Epub 2017 Oct 23. PMID 29089145
- [Background] Linardon J, Wade TD, de la Piedad Garcia X, Brennan L. The efficacy of cognitive-behavioral therapy for eating disorders: A systematic review and meta-analysis. J Consult Clin Psychol. 2017 Nov;85(11):1080-1094. doi: 10.1037/ccp0000245. PMID 29083223
- [Background] Linardon J, Wade TD. How many individuals achieve symptom abstinence following psychological treatments for bulimia nervosa? A meta-analytic review. Int J Eat Disord. 2018 Apr;51(4):287-294. doi: 10.1002/eat.22838. Epub 2018 Feb 8. PMID 29417609
- [Background] Masheb RM, Chan SH, Raffa SD, Ackermann R, Damschroder LJ, Estabrooks PA, Evans-Hudnall G, Evans NC, Histon T, Littman AJ, Moin T, Nelson KM, Pagoto S, Pronk NP, Tate DF, Goldstein MG. State of the art conference on weight management in VA: Policy and research recommendations for advancing behavioral interventions. J Gen Intern Med. 2017 Apr;32(Suppl 1):74-78. doi: 10.1007/s11606-016-3965-y. PMID 28271431
- [Background] Masheb RM, Grilo CM, Rolls BJ. A randomized controlled trial for obesity and binge eating disorder: low-energy-density dietary counseling and cognitive-behavioral therapy. Behav Res Ther. 2011 Dec;49(12):821-9. doi: 10.1016/j.brat.2011.09.006. Epub 2011 Sep 28. PMID 22005587
- [Background] Masheb RM, Lutes LD, Kim HM, Holleman RG, Goodrich DE, Janney CA, Kirsh S, Richardson CR, Damschroder LJ. High-frequency binge eating predicts weight gain among veterans receiving behavioral weight loss treatments. Obesity (Silver Spring). 2015 Jan;23(1):54-61. doi: 10.1002/oby.20931. Epub 2014 Nov 11. PMID 25385705
- [Background] Moss TP, Rosser BA. The moderated relationship of appearance valence on appearance self consciousness: development and testing of new measures of appearance schema components. PLoS One. 2012;7(11):e50605. doi: 10.1371/journal.pone.0050605. Epub 2012 Nov 30. PMID 23226326
- [Background] Phimphasone-Brady P, Dorflinger LM, Ruser C, Bullock A, Godfrey KM, Hernandez D, Min KM, Masheb RM. Self-report versus objective measurement of weight history: implications for pre-treatment weight gain. J Behav Med. 2019 Dec;42(6):1142-1147. doi: 10.1007/s10865-019-00045-0. Epub 2019 Apr 23. PMID 31016640
- [Background] Rosenberg, M. (1979). Conceiving the Self. New York: Basic Books.
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Sayer NA, Friedemann-Sanchez G, Spoont M, Murdoch M, Parker LE, Chiros C, Rosenheck R. A qualitative study of determinants of PTSD treatment initiation in veterans. Psychiatry. 2009 Fall;72(3):238-55. doi: 10.1521/psyc.2009.72.3.238. PMID 19821647
- [Background] Selim AJ, Rogers W, Fleishman JA, Qian SX, Fincke BG, Rothendler JA, Kazis LE. Updated U.S. population standard for the Veterans RAND 12-item Health Survey (VR-12). Qual Life Res. 2009 Feb;18(1):43-52. doi: 10.1007/s11136-008-9418-2. Epub 2008 Dec 3. PMID 19051059
- [Background] Sysko R, Walsh BT, Fairburn CG. Eating Disorder Examination-Questionnaire as a measure of change in patients with bulimia nervosa. Int J Eat Disord. 2005 Mar;37(2):100-6. doi: 10.1002/eat.20078. PMID 15732070
- [Background] Spielberger, C. D., Gorsuch, R. L., & Lushene, R. E. (1970). Manual for the State-Trait Anxiety Inventory. Polo Alto, CA: Consulting Psychologists Press.
- [Background] Spitzer RL, Yanovski S, Wadden T, Wing R, Marcus MD, Stunkard A, Devlin M, Mitchell J, Hasin D, Horne RL. Binge eating disorder: its further validation in a multisite study. Int J Eat Disord. 1993 Mar;13(2):137-53. PMID 8477283
- [Background] Joint Commission on Hospital Accreditation. APPROVED: New Requirements for Residential and Outpatient Eating Disorders Programs. Effective July 1, 2016, for Behavioral Health Care Accreditation Program. Jt Comm Perspect. 2016 Jan;36(1):4-9. No abstract available. PMID 26852462
- [Background] Udo T, Bitley S, Grilo CM. Suicide attempts in US adults with lifetime DSM-5 eating disorders. BMC Med. 2019 Jun 25;17(1):120. doi: 10.1186/s12916-019-1352-3. PMID 31234891
- [Background] Wilfley DE, Welch RR, Stein RI, Spurrell EB, Cohen LR, Saelens BE, Dounchis JZ, Frank MA, Wiseman CV, Matt GE. A randomized comparison of group cognitive-behavioral therapy and group interpersonal psychotherapy for the treatment of overweight individuals with binge-eating disorder. Arch Gen Psychiatry. 2002 Aug;59(8):713-21. doi: 10.1001/archpsyc.59.8.713. PMID 12150647
- [Background] Wilson GT, Wilfley DE, Agras WS, Bryson SW. Psychological treatments of binge eating disorder. Arch Gen Psychiatry. 2010 Jan;67(1):94-101. doi: 10.1001/archgenpsychiatry.2009.170. PMID 20048227
- [Background] Gusi, N., Olivares, P. R., & Rajendram, R. (2010). The EQ-5D health-related quality of life questionnaire. Handbook of Disease Burdens and Quality of Life Measures, 87-99.

DOCUMENTS (1):
  • Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT05304104/ICF_001.pdf